CLINICAL TRIAL: NCT06999772
Title: Combining Non-invasive Brain Stimulation and Physiotherapy to Improve the Management of Chronic Low Back Pain in Veterans
Brief Title: Combining Brain Stimulation and Physiotherapy for the Management of Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Chronic Pain Centre of Excellence for Canadian Veterans (Unknown); Foundation for Physical Medicine and Rehabilitation (Other)
Responsible Party: Principal Investigator, Hugo Massé-Alarie, Associate Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-3215 : DLPFC - PiP
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low-back Pain (cLBP)
Keywords: Non-invasive brain stimulation; comorbid psychological risk factors; chronic pain; repetitive transcranial magnetic stimulation; physiotherapy; pyschologically-informed; veterans
MeSH Terms: conditions — Chronic Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This is a single-blind, parallel-group, monocentric, randomised controlled trial (RCT).
Who Masked: Participant, Care Provider
Masking Description: The masking depends on the intervention:
  For rTMS, participants, treating physiotherapists and the statistician will be blinded to the group allocation. It is not possible to blind the rTMS technician because they need to choose the right TMS coil and muscle twitches in the face is elicited by the active rTMS.
  For physiotherapy, it is only possible to blind the statistician.
  Although the outcomes assessors are not blinded per se, the use of REDcap limits the possibility of bias related to outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active rTMS + PiP (Experimental): For weeks 1 and 2, participants will attend 5 brain stimulation sessions. During the first phase, the session will last 30-40 min (10-20 min of installation + 20 minutes of stimulation).
  In the second phase (weeks 3-8), brain stimulation and physiotherapy will be delivered in 2 separate sessions during the same week for 6 weeks. Each brain stimulation session will last 30-40 min and each physiotherapy session will last 30-45 min. Overall, participants will receive 11 sessions of rTMS only and 6 PiP sessions.
  Interventions: Device: Active rTMS; Other: Psychologically-informed physiotherapy (PiP)
- Sham rTMS + PiP (Sham Comparator): For weeks 1 and 2, participants will attend 5 sham brain stimulation sessions. During the first phase, the session will last 30-40 min (10-20 min of installation + 20 minutes of stimulation). In the second phase (weeks 3-8), brain stimulation and physiotherapy session will be delivered in 2 separate sessions during the same week for 6 weeks. Each sham brain stimulation session will last 30-40 min and each physiotherapy will last 30-45 min. Overall, participants will receive 11 sessions of sham rTMS only and 6 PiP sessions.
  Interventions: Device: Sham rTMS; Other: Psychologically-informed physiotherapy (PiP)
- Usual physiotherapy (Active Comparator): Participants will attend 6 sessions within 8 weeks (1session /week for 4 weeks, 1 session every 2 weeks between weeks 5-8). Each physiotherapy will last 30-45 min.
  Interventions: Other: Usual physiotherapy

INTERVENTIONS:
Device: Active rTMS — A figure-of-8 coil connected to a biphasic Magstim Rapid 2 stimulator (The MagstimCo, Whitland, UK) will be used. Coil orientation and position will be guided throughout the experiment by a neuronavigation system (Brainsight, Rogue research, Montreal, QC, Canada). Stimulation parameters will be obtained by measuring the motor threshold of the first right interosseous muscle, then the rTMS intensity will be set at 110% of this motor threshold. High frequency (HF) rTMS consisting of 60 trains of 5 s at 10 Hz with 15 s intertrain intervals, for a total of 3000 pulses per session, will be used. The coil will be positioned over the left dorsolateral PFC using the BeamF3 methods.
  Other Names: Repetitive Transcranial Magnetic Stimulation
  Arms: Active rTMS + PiP
Device: Sham rTMS — A sham coil will be used (e.g. equipped with a magnetic shield that blocks the magnetic field). The sham stimulation will last the same duration as the active rTMS and will be located over the same area (dorso-lateral prefrontal cortex).
  Other Names: Sham Repetitive Transcranial Magnetic Stimulation
  Arms: Sham rTMS + PiP
Other: Psychologically-informed physiotherapy (PiP) — Participants will receive 6 intervention sessions (45 min) over 6 weeks by a physiotherapist. The objective of this intervention is to identify biopsychosocial factors that may impede recovery and to address these factors within the physiotherapist's scope of practice. Physiotherapists will use strategies such as the establishment of common goals and therapeutic alliance, the use of behavior change model, motivational interview, education on pain neurophysiology, gradual exposure to movement and stress management strategies (e.g. breathing techniques). Participants allocated to PiP groups will have access to a website offering support information related to understanding their pain (e.g. pain neuroscience education), myths and false beliefs related to back pain, understanding the impact of psychological factors on their pain, self-management strategies, and healthy lifestyle habits. This site will be freely available to participants during the course of the study.
  Arms: Active rTMS + PiP; Sham rTMS + PiP
Other: Usual physiotherapy — Participants will receive 6 intervention sessions (45 min) over 8 weeks by a physiotherapist. This is a pragmatic group that aims to represent real-word clinical practice i.e. interventions commonly used in physiotherapy to manage CLBP. All interventions that a physiotherapist can deliver in the province of Quebec will be allowed (e.g. manual therapy, exercises). No training will be provided to better reflect usual clinical practice in physiotherapy.
  Arms: Usual physiotherapy

SUMMARY:
Chronic low back pain (CLBP) is a major health challenge in Canada, leading to substantial disability and socioeconomic burden, particularly among Veterans. In military Veterans, LBP is the most common chronic pain condition. Conventional interventions have limited effectiveness. The refractoriness to interventions suggests that specific CLBP mechanisms may be missed by current treatments, prompting a shift towards psychologically informed approaches which aim to address emotional and cognitive factors alongside biomedical aspects. The integration of these concepts into physiotherapy is called psychologically informed physiotherapy (PiP). Despite promising results of PiP from randomized controlled trials, residual pain and disability often persist in Veterans. Non-invasive brain stimulation, such as repetitive transcranial magnetic stimulation (rTMS), may enhance the effectiveness of PiP by modulating cognition, emotion, and pain. This proposal seeks to determine whether non-invasive brain stimulation can enhance the effects of PiP.

DETAILED DESCRIPTION:
The study will compare the effects of (1) combining rTMS with PiP, (2) PiP alone (+sham rTMS), and (3) usual physiotherapy (UP) on physical functioning in Veterans suffering from CLBP and comorbid psychological factors associated with back pain. Participants will undergo an 8-week intervention program. Validated questionnaires will be used to measure outcomes at baseline, 2-, 8-, and 26-week follow-ups. The main objective is to determine if the combination of PiP and rTMS is superior to PiP and UP alone to improve physical functioning in Veterans suffering from CLBP and comorbid psychological factors.

The secondary objectives are to compare the effectiveness of these interventions on secondary outcomes, that are, pain intensity, quality of life, movement pain-related fear, pain catastrophizing, self-efficacy, depression symptoms, medication use and post-traumatic stress disorder symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 65 years old
* Military Veterans with non-specific chronic low back pain (> 3 months, > 50% of the days in the last 6 months)
* High level of psychosocial factors, scoring ≥4 on the Start Back Screening Tool
* Functional limitations, scoring ≥ 15% on the Oswestry Disability Index (ODI)

Exclusion Criteria:

* Non-musculoskeletal conditions causing low back pain (e.g., neoplasia, fracture)
* Diagnosis of drug or alcohol abuse
* Change of drug dosage in the last month for the treatment of pain or mental health
* Presenting with any specific rTMS-related exclusion criteria such as previous seizure/convulsion, cochlear implant, and pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Physical functioning (ODI) | Baseline, weeks 2, 8 and 26.
  The Oswestry Disability Index (ODI) is a self-completed questionnaire on estimated disability including 10 questions rated on a 6-item scale, from 0 (no disability) to 5 points (maximal disability). The total score ranges from 0 (no disability) to 100% (maximal disability).

SECONDARY OUTCOMES:
Pain intensity (NPRS) | Baseline, weeks 2, 8 and 26.
  The Numerical Pain Rating Scale (NPRS) is an 11-point scale used to measure the mean intensity of pain in the last week ranging from 0 (no pain) to 10 (worst imaginable pain).
Quality of life (EQ-5D-5L) | Baseline, weeks 2, 8 and 26.
  The EQ-5D-5L is a self-administrated questionnaire that contains 5 questions, each rated on a 5-point scale and mesuring 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. These dimensions define 5^5 = 3125 possible health states, which can be converted into a Canadian weighted index score. This index score ranges from -0.148 (lowest value assigned to a health state) to 0.949 (highest value assigned to a health state).
Depression symptoms (PHQ) | Baseline, weeks 2, 8 and 26.
  The Patient Health Questionnaire is a self-administrated questionnaire of 9 questions used to diagnose depression and grade severity of symptoms. The scale ranges from 0 to 27; a higher score means more depressive symptoms.
Pain catastrophizing (PCS) | Baseline, weeks 2, 8 and 26.
  The Pain Catastrophizing Scale (PCS) is a self-administrated questionnaire of 13 questions measuring catastrophizing thoughts contributing to pain on a 5-point scale ranging from 0 (not at all, low level of catastrophizing thoughts) to 5 (all the time, high level of catastrophizing thoughts).
Fear of movement (TSK-13) | Baseline, weeks 2, 8 and 26
  The Tampa Scale of Kinesiophobia is a self-administrated questionnaire used to assess fear of movement using 13 questions on a 4-point scale ranging from 1 (strongly disagree, low level of kinesiophobia) to 4 (strongly agree, high level of kinesiophobia).
Self-efficacy (PSEQ-10) | Baseline, weeks 2, 8 and 26.
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questionnaire mesuring the confidence people with ongoing pain have in performing activities while in pain, on a 10-point scale from 0 (not at all confident, low self-efficacy) to 10 (completely confident, high self-efficacy).
Post-traumatic stress disorder (PCL-5) | Baseline, weeks 2, 8 and 26.
  The Posttraumatic Stress Disorder Checklist (PCL-5) is a 20-item self-completed questionnaire that assesses the 20 DSM-5 symptoms of post-traumatic stress disorder on a 5-point scale ranging from 0 (not a all, no symptoms of PTSD) to 4 (extremely, severe symptoms of PTSD).
Medication use | Baseline, weeks 2, 8 and 26.
  The Medication Quantification Scale Version 4 quantifies the risk weights of the use of 36 drug sub-classes used in pain management. Each drug sub-class has a detriment weight from 0 (low risk weight) to 10(high risk weight). The total score represents the summation of each drug class used by the participant.
Global rating of change (GRC) | Weeks 2, 8 and 26
  The Global rating of change (GRC) is a 11-point scale ranging from -5 (a great deal worst) to 5 (a great deal better) to measure the perceived change of health status after the intervention.
Patient Acceptable Symptom State (PASS) | Baseline, weeks 2, 8 and 26.
  The Patient Acceptable Symptom State (PASS) measures if the participants consider their current functional and symptoms states as satisfactory or not. A visual analogue scale ranging from 0 (completely dissatisfied) to 100 (completely satsified) is used.

OTHER OUTCOMES:
Adverse events | Weeks 2, and 8
  All adverse events and reasons for drop-out will be recorded and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Massé-Alarie, PhD, Principal Investigator — Laval University
Locations (2):
- Canada (2):
  - Centre interdisciplinaire de recherche en réadaptation et intégration sociale (CIRRIS), Québec, Quebec
  - Cirris (Centre Interdisciplinaire de Recherche en Réadaptation et Intégration Sociale), Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (IPD) that underlie the results reported in the published article will be made available. The study protocol will also be published.
Supporting Information: Study Protocol
Time Frame: Data will become accessible after the publication and will remain accessible for a period of 5 years after initial release.
Access Criteria: Access to IPD will be granted to qualified researchers whose proposals are methodologically sound and ethically approved. Researchers must obtain approval from their Institutional Review Board (IRB), Research Ethics Board (REB), or equivalent ethics committee, and must sign a Data Use Agreement (DUA) before receiving any data.
  Requests for access should be submitted to: hugo.masse-alarie@fmed.ulaval.ca.

REFERENCES:
- [Derived] Dupuis F, Tousignant-Laflamme Y, Marier Deschenes P, Fournier P, Nduwimana I, Ballot O, Loisel L, Pinard AM, Lacombe L, Langevin P, Gaumond A, Roy JS, Masse-Alarie H. Combining Noninvasive Brain Stimulation and Physiotherapy to Improve the Management of Chronic Low Back Pain in Veterans: Protocol for a Multi-Arm Randomized Controlled Trial. JMIR Res Protoc. 2026 Jan 26;15:e78952. doi: 10.2196/78952. PMID 41587077